CLINICAL TRIAL: NCT02967952
Title: A RCT on Supraglottic Airway Versus Endotracheal Intubation in OHCA (SAVE)
Brief Title: A RCT on Supraglottic Airway Versus Endotracheal Intubation in OHCA
Acronym: SAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201606047RINA
Record Dates: First submitted 2016-10-20; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Prehospital Airway Management in Patients With Cardiac Arrest
Keywords: out-of-hospital cardiac arrest (OHCA); supraglottic airway (SGA); endotracheal intubation (ETI); emergency medical system (EMS); Supraglottic Airway Versus Endotracheal tube (SAVE)
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- supraglottic airway (SGA) (Active Comparator): Adult patients with non-trauma causes of OHCA who are resuscitated by emergency medical technician paramedic (EMTP) in the prehospital setting and received airway management of supraglottic airway (SGA).
  Interventions: Device: supraglottic airway (SGA) V.S. endotracheal intubation (ETI)
- endotracheal intubation (ETI) (Active Comparator): Adult patients with non-trauma causes of OHCA who are resuscitated by emergency medical technician paramedic (EMTP) in the prehospital setting and received airway management of endotracheal intubation (ETI).
  Interventions: Device: supraglottic airway (SGA) V.S. endotracheal intubation (ETI)

INTERVENTIONS:
Device: supraglottic airway (SGA) V.S. endotracheal intubation (ETI) — already being described above

SUMMARY:
In this 3-year successive research plan, investigators will conduct a prehospital randomized controlled trial to address the following question: In adult patients with non-traumatic cause of out-of-hospital cardiac arrest resuscitated by emergency medical technician (paramedic level) in the prehospital setting, will receiving endotracheal tube intubation cause a better chance of sustained recovery of spontaneous circulation and other survival outcomes like neurologically favorable status, comparing to those who receiving supraglottic airway device.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest; OHCA
* age ≥ 20 years old
* non-traumatic cause

Exclusion Criteria:

* signs of obvious death, eg. decapitation or rigor mortis
* theoretically not suitable for ETI, eg. facial deformity or third-trimester pregnancy
* theoretically not suitable for SGA, eg. foreign-body airway obstruction
* with "do not attempt resuscitation" order
* the occurrence of OHCA during ambulance transport
* ROSC in the field with clear consciousness and spontaneous adequate ventilation
* advanced airway being established before the arrival of paramedics

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
survival to admission | One month after event
  Measurement of outcome by standard Utstein OHCA registry system in Taipei City

SECONDARY OUTCOMES:
any ROSC | One month after event
  Measurement of outcome by standard Utstein OHCA registry system in Taipei City
survival to discharge | One month after event
  Measurement of outcome by standard Utstein OHCA registry system in Taipei City
favorable neurologic outcome | One month after event
  Favorable neurologic outcome was defined by CPC (cerebral performance category) 1 and 2.
  Measurement of outcome by standard Utstein OHCA registry system in Taipei City

OTHER OUTCOMES:
The rate of survival to discharge of OHCAs resuscitated by non-paramedic (airway device: all SGA) | One month after event
  Measurement of outcome by standard Utstein OHCA registry system in Taipei City
The interaction between age and airway management | One month after event
  Deciphering interactions in logistic regression model with variables of standard Utstein OHCA registry system in Taipei City
The interaction between bystander CPR and airway management | One month after event
  Deciphering interactions in logistic regression model with variables of standard Utstein OHCA registry system in Taipei City
The interaction between shockable rhythms and airway management | One month after event
  Deciphering interactions in logistic regression model with variables of standard Utstein OHCA registry system in Taipei City

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chu Chiang, MD, PhD., Principal Investigator — Emergency Dept, National Taiwan University Hospital

REFERENCES:
- [Derived] Lee AF, Chien YC, Lee BC, Yang WS, Wang YC, Lin HY, Huang EP, Chong KM, Sun JT, Huei-Ming M, Hsieh MJ, Chiang WC. Effect of Placement of a Supraglottic Airway Device vs Endotracheal Intubation on Return of Spontaneous Circulation in Adults With Out-of-Hospital Cardiac Arrest in Taipei, Taiwan: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2148871. doi: 10.1001/jamanetworkopen.2021.48871. PMID 35179588